CLINICAL TRIAL: NCT01560806
Title: Quasi-experimental Intervention Study on Hypertension Management Combined With Comprehensive Healthy Lifestyle Promotion at Commune Level
Brief Title: Intervention Study on Hypertension Management Combined With Health Promotion at Commune Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National Heart Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VNHI-07-001
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Hypertension; Cardiovascular Risk Factor; Lifestyle
Keywords: hypertension; cardiovascular risk factor; lifestyle
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Healthcare services (No Intervention): People with high blood pressure detected during screening survey or opportunistically during study period will be referred to receive the conventional health care services for hypertension at district hospital or local commune health station
- Commune Hypertension Management (Experimental): People with high blood pressure were managed in commune-based hypertension management programme
  Interventions: Other: Commune Hypertension Management

INTERVENTIONS:
Other: Commune Hypertension Management — People with high blood pressure will be invited to join the management programme, with monthly check-up, delivery of multi anti-hypertensive drugs and lifestyle consultation.
  Antihypertensive drugs delivered to local patients included (1) low-dose hypothiazide diuresis, (2) calcium channel blocker and (3) ACEI
  Other Names: Commune-based Hypertension Management
  Arms: Commune Hypertension Management

SUMMARY:
A quasi-experimental study design was chosen to compare the model of hypertension management at commune-level with conventional management for people with high blood pressure in two communes (one for intervention versus one for reference).

A intervention model included the commune-based programme on hypertension management combined with comprehensive health promotion campaigns

DETAILED DESCRIPTION:
A quasi-experimental study design was chosen: two communes were purposively selected from Ba-Vi setting: Phu-Phuong for reference and Phu-Cuong for intervention communes A hypertension management programme and the nested comprehensive health promotion campaigns were implemented simultaneously in Phu-Cuong while nothing performed in Phu-Phuong except for local conventional healthcare services.

The health promotion campaigns aimed at smoking cessation, reduction of alcohol consumption, encourage of unsalted diet and physical activity, all of which targeted to every local inhabitants.

The hypertension management programme focused on monthly check-ups, drug delivery and individual lifestyle consultation, all of which targeted to hypertensives only.

Baseline cross-sectional survey was used to assess cardiovascular pattern in local community before intervention and recruit people with high blood pressure for the management programme in intervention commune Repeated cross-sectional surveys were used to evaluate the impacts of health promotion.

Cohort study on hypertensives was used to evaluate the impacts of the management programme.

ELIGIBILITY:
Inclusion Criteria:

* Adult people above 25

Exclusion Criteria:

* People deny to join the study

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of people with high blood pressure receiving treatment and being controlled in intervention commune | Baseline and after 3-year
  Changes in proportion of treated and controlled hypertension after 3-years intervention compared to baseline

SECONDARY OUTCOMES:
Changes in prevalences of behavioral cardiovascular risk factors in intervention commune | Baseline and after 3-year
  Changes in prevalence of behavioral cardiovascular risk factors after 3-years intervention compared to baseline
Changes in average blood pressure in the population in intervention commune | Baseline and after 3 years
  Changes in average systolic and diastolic blood pressure in the studied population after 3-year intervention

CONTACTS AND LOCATIONS:
Overall Officials: Son T. Pham, MD, Principal Investigator — Vietnam National Heart Institute
Locations (1):
- Vietnam National Heart Institute, Hanoi, Hanoi, Vietnam

REFERENCES:
- See also: Information involved in the National Targeted Programme on Hypertension Prevention and Control — http://www.huyetap.vn